CLINICAL TRIAL: NCT03222700
Title: The Recovery Profiles After Robotic or Open Thyroidectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B-1606/351-005
Record Dates: First submitted 2017-07-12; First posted 2017-07-19 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Postoperative Sorethroat; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- robotic thyroidectomy group
  Interventions: Procedure: surgical procedure
- open thyroidectomy group
  Interventions: Procedure: surgical procedure

INTERVENTIONS:
Procedure: surgical procedure — In robotic thyroidectomy group, patients are received surgery using robotic system. In open thyroidectomy group, patients are received conventional open surgery.

SUMMARY:
In the present study, The investigators investigated the effect of surgical methods on the recovery of patients after robotic surgery and open thyroidectomy

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing robotic thyroidectomy or open conventional thyroidectomy
2. Adults 19 to 70 years of age
3. American Society of Anesthesiologists Physical grade 1-2

Exclusion Criteria:

1. Patients who underwent surgery on the neck and in the laryngeal area before
2. Patients who do not understand or can not express pain scale
3. Patients with sore throat and cough before surgery
4. If intubation is difficult or repeated intubation is performed
5. Patients who are using opioids or analgesics as chronic agents.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing robotic thyroidectomy or open conventional thyroidectomy
Sampling Method: Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
postoperative sore throat | postoperative 1 hour
  none, mild, moderate, severe

CONTACTS AND LOCATIONS:
Locations (1):
- Ah-young Oh, Seongnam-si, Gyeonggi-do, South Korea